CLINICAL TRIAL: NCT01557998
Title: Testing and Linkage to Care for IDUs in Kenya (TLC-IDU Kenya); HCV Among PWIDs in Kenya: A Supplement to the TLC-IDU Study
Brief Title: Testing and Linkage to Care for Injecting Drug Users in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: NYU Langone Health (Other); Kenya National AIDS & STI Control Programme (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1512016965; R01DA032080 (NIH); R01DA032080-05S1 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-03-20 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: HIV Infection; HCV Coinfection
Keywords: Test and linkage to care; Injecting drug user (IDU); Prevention with positives; ART adherence; point of care CD4 counts; Peer case management; Conditional cash transfer
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control - No intervention (Other): PWID in the control arm will receive the behavioral survey, follow-up interviews, health education and training sessions on how to recruit peers, the rapid HIV and HCV test, and the point of care CD4 test but will not be assigned a peer case manager. Confirmed HCV viremic will receive HCV treatment.
  Interventions: Drug: HCV+PWID; Behavioral: Control - No intervention
- POC CD4 and Peer Case Management (Experimental): HIV-positives will receive prevention with positives (PwP) counseling and point of care CD4 counts. Those with CD4 <500/μL will be assigned a peer case manager to link the person to ART at study-participating HIV clinics, support ART and PwP adherence and care retention. Confirmed HCV viremic will receive HCV treatment.
  Interventions: Behavioral: POC CD4 and Peer Case Management; Drug: HCV+PWID
- HCV+PWID (Other): Control and Experimental Confirmed HCV viremic study subject will receive HCV treatment
  Interventions: Drug: HCV+PWID

INTERVENTIONS:
Behavioral: POC CD4 and Peer Case Management — HIV-positives will receive prevention with positives (PwP) counseling and point of care CD4 counts. Those with CD4 <500/μL will be assigned a peer case manager to link the person to ART at study-participating HIV clinics, support ART and PwP adherence and care retention.
  Arms: POC CD4 and Peer Case Management
Drug: HCV+PWID — Deliver direct acting antiviral (DAA) regimens for HCV+PWID. We will treat both active and inactive confirmed HCV viremic PWID from either Medication Assisted Treatment (MAT) clinics in Nairobi, Mombasa, and Malindi, Kenya or Collaborating partners' sites/Drop-in Centers (DICs) in Mombasa and Mtwapa, Kenya with direct acting antiviral (DAA) regimens. The mode of treatment delivery will be Directly Observed Therapy (DOT) for 84 consecutive doses (one dose per day). All participants will receive pre, post and ongoing counseling as per study protocol.
  Other Names: Deliver ongoing counseling
Behavioral: Control - No intervention
  Arms: Control - No intervention

SUMMARY:
Testing and Linkage to Care for Injecting Drug Users in Kenya:

Interventions for people who inject drugs (PWID) in sub-Saharan African have been almost entirely absent, despite the fact that in countries like Kenya they contribute a growing proportion of incident HIV infections. This study will leverage a historic decision in Kenya to launch needle exchange program (NSP) and related services for this most-at-risk population (MARP). The investigators will use this NSP/MARP platform to seek out PWID, deliver rapid HIV testing, point of care CD4 count and link to ART using peer case managers, and evaluate community viral load impact using a stepped wedge cluster-randomized design. Lessons learned will have important applicability throughout sub-Saharan African.

HCV Among PWID in Kenya: A Supplement to the TLC-IDU study:

The prevalence of HCV in Kenya, where an increasing number of people who inject drugs (PWID) live and are becoming HIV- as well as HCV-infected, has not been defined. We will establish HCV prevalence among PWID in Nairobi, Western, and Coastal region by adding HCV rapid and confirmatory tests in our parent PWID study (TLC-IDU Kenya); deliver appropriate counseling and treatment options to those eligible; collect HCV treatment adherence data; and disseminate study findings. These data will provide novel and relevant information about HCV and HIV co-infection in Kenya among PWID that will be immediately applicable in terms of public health impact to national and regional HCV testing, counseling, and clinical management policy.

DETAILED DESCRIPTION:
Testing and Linkage to Care for Injecting Drug Users in Kenya

The purpose of the study will be to leverage the GoK's first-ever needle and syringe program, to implement the HIV seek, test, treat, and retain paradigm among PWID, whose parenteral and sexual transmission networks amplify HIV epidemics. Study innovations include: (1) use of a stepped wedge trial design; (2) intent to track community viral load in a low-income country setting; (3) use of rapid CD4 assays to reduce time from HIV diagnosis to ART initiation; and (4) use of conditional cash transfers to support peer case management of participant HIV treatment retention.

Aim 1: Evaluate seek test treat retain using a stepped wedge cluster-randomized design. Clusters will be the planned NSP service sites. The investigators will initiate respondent-driven sampling (RDS) to reach PWID in Nairobi, Western region and coastal Mombasa (including Malindi) for baseline HIV-1 prevalence determination, then collect waves of study data as service sites roll out, including behavioral data. Teams will do rapid HIV and HCV testing and refer for addiction/mental health and other services (e.g., OST). HIV-positives will receive prevention with positives (PwP) counseling and point of care CD4 counts. Those with CD4 <500/μL will be assigned a peer case manager to link the person to ART at study-participating HIV clinics, support ART and PwP adherence and care retention. Both peer case managers and subjects will receive small conditional cash transfers for subject's adherence to HIV care visits. Primary study outcomes will include time to successful linkage to care, time to ART, and community viral load before and after TLC-IDU initiation. 'Community viral load' will be ascertained by collecting specimens from randomly-selected HIV-positives at each of the NASCOP NSP-IDU service sites. This sampling will be done in waves over time, to document changes in infectivity (median viral load). With individual viral loads collected per site per time step (for a n= of at least 1800 viral loads in total across all sites and timewaves) the investigators will have good power to detect log10 viral load changes of 0.23 and hazard ratios of ~1.5 when comparing pre- and post-intervention period using linear mixed effects analysis.

Aim 1: Research hypothesis: Staggered rollout of a planned NSP/MARP program can be utilized to collect pre- and post intervention data that will allow assessment of impact on community viral load. Linkage to care will be higher, time to ART initiation will be reduced, and retention in care will be higher during time periods with the TLC-IDU services as compared to time periods with standard of care.

Aim 2: Conduct mathematical modeling to estimate community viral load in PWID injecting and sexual networks, and to assess potential population-level impact of the TLC-IDU intervention on Ro, numbers of infections averted, and quality-adjusted life expectancy.

Aim 2: Research hypothesis: HIV transmission dynamics models can use parameters from Aim 1 data waves, with sensitivity analyses identifying those parameters with largest impact on effect estimation and stability.

Aim 3: Assess the incremental cost-effectiveness ratio of the TLC-IDU model, using a national payer perspective. This study will provide among the world's first data regarding implementation of the seek, test, treat and retain paradigm with IDUs in sub-Saharan Africa. It will demonstrate the degree to which a combination of structural, biomedical and behavioral interventions can reduce infectivity. Partnership with Kenya's national HIV program will allow lessons learned from this study to inform other countries considering how best to address the growing PWID contribution to the HIV epidemic in this high-HIV-burden region.

Aim 3: Research hypothesis: Utilizing MARP/NSP services will result in a reduction in median community viral load and in forward HIV transmission. Cost per quality adjusted life year saved and HIV infection averted will be favorable as compared with the alternative of no specific seek, test, treat and retain program directed to PWID.

HCV Among PWID in Kenya: A Supplement to the TLC-IDU study

Hepatitis C virus (HCV) is a global pandemic that leads to 500,000 preventable deaths worldwide. People who inject drugs (PWID) are at much higher risk of HCV infection, with an estimated 10 million HCV infections among PWID worldwide. In Kenya, PWID are at high risk of HCV infection, yet HCV prevalence in this key population is not well-defined. The time is ripe to establish HCV prevalence among high-risk PWID in Kenya, determine the role of sexual transmission and risk behavior in those identified with HCV, and explore potential best approaches to provide clinical and counseling services, especially to HCV-HIV co-infected individuals. We therefore propose to add rapid HCV testing to our study of PWID in Kenya, the NIDA-funded parent 'TLC-IDU study' (Kurth & Cherutich, PIs), and to collect additional specific behavioral and clinical data relevant to HCV in this high-HIV burden setting.

These data will provide novel and highly relevant information about HCV and HIV co-infection in Kenya among PWID that will be immediately applicable to national HCV testing and treating policy. Our scientific objectives:

Supplement Specific Aim 1: Establish HCV prevalence in PWID in Nairobi, Western and Coastal region, by adding a rapid HCV assay to the study panel among all participants (both HIV infected and uninfected) recruited during the last TLC-IDU study waves. (The study involves recruiting PWID who undergo rapid HIV testing/phenotyping and behavioral data collection, as well as peer case management to support HIV treatment). Those testing positive with the HCV rapid point of care assay will be given initial counseling to raise their awareness, tell them they have been exposed, and encourage them to return for confirmatory results. Confirmatory viral HCV testing will be done and confirmed positive participants given an incentive to return to the study site for standardized HCV counseling and treatment referral for those with HCV monoinfection and HIV-HCV infection. Main outcomes will include: a) HCV prevalence determination b) HCV testing and counseling feasibility and acceptability measures, c) unique predictors of HCV monoinfection and HIV and HCV coinfection determined in multinomial logistic regression analysis.

Supplement Specific Aim 2: Deliver HCV counseling and available treatment, including sofosbuvir treatment to those eligible and collect HCV treatment adherence data.

Supplement Specific Aim 3: Present study findings and program implications at a national workshop with study partner NASCOP. Invite key stakeholders, researchers, and implementers to discuss HCV agenda for Kenya.

ELIGIBILITY:
The intervention phase with stepped wedge rollout of TLC-IDU-MARP sites Inclusion Criteria:

* subjects will be adults (≥18 year olds)
* attend NSP/MARP service sites
* live in Nairobi (Central Province), Western region, or coastal Mombasa (Coast Province including Malindi), Kenya
* are IDUs that ever injected any non-prescribed drugs
* are IDUs that have used any non-prescribed drugs within the past 12 months
* for HIV viral load testing, individuals must have tested HIV+
* for HCV viral load testing, individuals must have been confirmed HCV viremic

Exclusion Criteria:

* subjects are not adults (<18 years old)
* do not attend NSP/MRP sites
* do not live in Nairobi (Central Province), Western region, or coastal Mombasa (Coast Province including Malindi), Kenya
* are not IDUs
* for viral load testing, individuals who tested HIV-
* for HCV viral load testing, individuals who were confirmed HCV NOT viremic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9449 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Linkage to care and time to ART | Data collection done in 5 waves separated by 6 months
  Use of rapid CD4 assays to reduce time from HIV diagnosis to ART initiation
Community viral load before and after the TLC-IDU initiation | Data collection done in 5 waves separated by 6 months
  Community viral load will be ascertained by collecting specimens from randomly-selected HIV-positives at each of the NASCOP NSP-IDU service sites. This sampling will be done in waves over time, to document changes in infectivity (median viral load).
Retention in Care | Data collection done in 5 waves separated by 6 months
  HIV-positives will receive prevention with positives (PwP) counseling and point of care CD4 counts. Those with CD4 <500/μL will be assigned a peer case manager to link the person to ART at study-participating HIV clinics, support ART and PwP adherence and care retention.
HCV prevalence determination | Data collection done in wave 6 - 6-month-period
  Establish HCV prevalence in PWIDs in Nairobi, Western and Coastal region, by adding a rapid HCV assay to the study panel among all participants (both HIV infected and uninfected) recruited during the last TLC-IDU study waves
HCV testing and counseling feasibility and acceptability measures | Done in wave 6 - 6-month-period
  Offering HCV testing and counseling to all study participants. Offering treatment referral for those with HCV monoinfection and HIV-HCV infection

SECONDARY OUTCOMES:
Modeling HIV transmission dynamics | End of study (will occur in year 5 of the study)
  Conduct mathematical modeling to estimate community viral load in PWID injecting and sexual networks, and to assess potential population-level impact of the TLC-IDU intervention on Ro, numbers of infections averted, and quality-adjusted life expectancy.
Assess the incremental cost-effectiveness ratio of the TLC-IDU model | End of study (will occur in year 5 of the study)
  The expectation is that utilizing MARP/NSP services will result in a reduction in median community viral load and in forward HIV transmission. Cost per quality adjusted life year saved and HIV infection averted will be favorable as compared with the alternative of no specific seek, test, treat and retain program directed to IDUs.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kurth, PhD, CNM, Principal Investigator — Yale University School of Nursing; Peter Cherutich, MD, PhD, MPH, Principal Investigator — NASCOP, MoH Kenya
Locations (1):
- National AIDS/STD Control Programme (NASCOP), Nairobi, Kenya